CLINICAL TRIAL: NCT06227780
Title: FX ENTRAIN: Perturbation of Neurodynamics Underlying Sensory Hyperarousal and Statistical Learning in Youth With FXS
Brief Title: Alpha Auditory Entrainment for Cognitive Enhancement and Sensory Hypersensitivity in Youth With Developmental Disorders
Acronym: ENTRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ernest Pedapati, MD, Assistant Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-0911; 1R01HD108222-01 (NIH)
Record Dates: First submitted 2023-11-16; First posted 2024-01-29 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Fragile X Syndrome; Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome
Keywords: Neurodevelopmental Disorders; Autistic Disorder; Autism Spectrum Disorder; Fragile X Syndrome; Fragile X; FXS; ASD; Asperger; Autism
MeSH Terms: conditions — Fragile X Syndrome; Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Neurodevelopmental Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: All visits across all arms will follow identical procedures. Aim 1 and Aim 2 consist of a case-control study that will be completed over two visits, in which baseline data will be collected from participants that will be used to optimize the intervention delivered in Aim 3. Aim 3 consists of a two-visit, randomized controlled, crossover acute perturbation study to study the effect of alpha auditory entrainment (AAE) or sham stimulation on brain activity. AAE will be performed in two visits as a double-blind, sham-controlled crossover study such that each participant will receive AAE and sham in random order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As the randomization and "dispensing" of the intervention is conducted via software, investigators, study staff, and study subjects will all be blinded to the randomized study treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fragile X Syndrome (Experimental): Fragile X Syndrome with full FMR1 mutations (>200 CGG repeats; at least partial FMR1 gene methylation)
  Interventions: Other: Alpha Auditory Entrainment; Other: Sham
- Autism Spectrum Disorder Controls (Active Comparator): Age and sex-matched with FXS cohort
  Interventions: Other: Alpha Auditory Entrainment; Other: Sham
- Typically Developing Controls (Active Comparator): Subjects with neither disorder who have met normal developmental milestones
  Interventions: Other: Alpha Auditory Entrainment; Other: Sham

INTERVENTIONS:
Other: Alpha Auditory Entrainment — Alpha Brainwave Entrainment (AAE) stimulus: starts at high theta range (7-Hz) through high alpha (13-Hz) in 2 Hz steps on a 500 Hz sine carrier tone
  Target frequency: 10 Hz
  Delivery: headphones/speakers
  Other Names: Alpha Brainwave Entrainment; Alpha Binaural Beats; Pulsed Sound Stimulation; Sonic Entrainment
Other: Sham — Sham stimulus: carrier tone alone
  Target frequency: N/A
  Delivery: headphones/speakers

SUMMARY:
Fragile X Syndrome (FXS) is a complex neurodevelopmental disorder caused by a mutation on the X chromosome. Scientists have investigated FXS extensively in both humans and animals. Thus far, phenotypic rescue in animal models has not resulted in treatment breakthroughs in humans, though some important discoveries have been made. Research has shown that individuals with FXS process sounds differently than those in the typical population, and they also show baseline differences in brain activity, including high gamma activity, increased theta activity, and decreased alpha activity. The investigators' central hypothesis is that these alterations in brain activity (specifically alpha and gamma activity) impair the brain's ability to process new information, thereby impeding cognitive functioning and increasing sensory sensitivity. The investigators propose that auditory entrainment, a technique that involves playing special sounds through headphones, will normalize brain activity in individuals with FXS and lead to increased cognitive function and decreased sensory hypersensitivity.

DETAILED DESCRIPTION:
Fragile X Syndrome (FXS) is an exemplar monogenetic neurodevelopmental disorder (NDD) where a tremendous body of multi-species translational research has elucidated the underlying molecular pathophysiology, and more recently, in-depth electrophysiology of cortical function. Thus far, phenotypic rescue in animal models has not resulted in treatment breakthroughs in humans. Central to this discrepancy is a poor understanding of the constituent neurodynamics of averaged group effects and individual variability in human brain activity as related to higher-level cognitive symptomatology and clinical phenotype. The investigators' large collection of preliminary data demonstrates that individuals with FXS do not mount precise neural responses to the sensory auditory chirp and, instead, have "noisy" asynchronous gamma activity. Furthermore, a marked reduction in alpha power suggests altered thalamocortical function, reducing the ability to detect signal from noise and representing potential tractable targets for "bottom-up" entrainment. This approach involves three scientific aims, which, if addressed, would ascertain underlying mechanisms that may alleviate sensory and cognitive impairments. First, the investigators will study transient, non-continuous features (neurodynamics) of alpha and gamma oscillations in resting-state EEG and sensory auditory chirp that model patient-level heterogeneity and constitute group effects (Aim 1A), and will also identify what, if any, of these novel features are conserved in the Fmr1-/-KO using preexisting murine EEG data and represent patient subgroups (Aim 1B). Second, the research team will extend into cognition by studying neurodynamics and circuit modeling associated with statistical learning (SL), which shares similar neural mechanisms to the sensory auditory chirp (Aim 2). Third, the investigators will use individualized closed-loop alpha auditory entrainment (AAE) to attempt the normalization of neural signatures of the sensory auditory chirp and SL tasks (Aim 3). Aim 1 and 2 findings will provide critical data to optimize closed-loop parameters of AAE to serve as a "bottom- up" neural probe to understand the mechanics of disorder-relevant circuit activity through perturbation of thalamocortical drive. Ascertaining the mechanisms underlying these alterations would have a high clinical impact, especially to enhance early intervention to alter the trajectory of intellectual development in which no definitive treatments are available.

ELIGIBILITY:
Inclusion Criteria:

* FXS Cohort: 1) Aged 5-10 years, inclusive; 2) Patient has full FMR1 mutation confirmed by genetic testing.
* ASD Cohort: 1) Aged 5-10 years, inclusive; 2) Have no known genetic mutation; 3) Have documentation of ASD diagnosis; 4) Score ≤ 15 on SCQ screen; 5) Be in good health per investigator.
* TDC Cohort: 1) Aged 5-10 years, inclusive; 2) Have no known genetic mutation; 3) Have documentation of ASD diagnosis; 4) Score ≤ 15 on SCQ screen; 5) Be in good health per investigator; 6) Patient has met normal developmental milestones; Patient has no family history of heritable neuropsychiatric disorders; 7) Patient has an IQ greater than 85 on the Stanford-Binet; 8) Score ≤8 on an SCQ screen.

Exclusion Criteria:

* All subjects: 1) Patient has auditory or visual impairments that cannot be corrected; 2) History of substance abuse or dependence within the past 6 months

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2028-05-24 (Estimated)

PRIMARY OUTCOMES:
Alpha auditory entrainment versus sham effect on Word Learning Index during the Statistical Learning Passive Task. | 1 week
  The Statistical Learning Passive Task uses an EEG-based measure of neural entrainment that uses inter-trial coherence (ITC) to calculate Word Learning Index (WLI).
  Patterns of EEG phase-locking, corresponding to a shift in processing from raw syllable units to cohesive words, reflect gradual statistical learning in the brain. The WLI effect can be quantified by creating a ratio of the inter-trail coherence for words versus syllables, as follows:
  WLI = Inter-trial Coherence word rate / Inter-trial Coherence syllable rate
  A higher WLI indicates a relatively stronger response to tri-syllabic nonwords compared to raw syllables, reflecting stronger word segmentation due to statistical learning.

OTHER OUTCOMES:
Alpha auditory entrainment versus sham effect on the Behavior Learning Effect during the Statistical Learning Active Task. | 1 week
  The Active SL Task based measure uses reaction time to estimate a behavioral measure of SL, the Behavioral Learning Effect BLE. BLE values indicate greater proportional facilitation to predictable words in the stream, indicative of stronger SL at the individual level. The Behavioral Learning effect is quantified as follows:
  BLE (in ms) = (Reaction time target syllable position 1)-(Reaction time target syllable position 3)
  Larger BLE values indicate greater proportional facilitation to predictable words in the stream, indicative of stronger SL at the individual level.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest V Pedapati, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
all collected, deidentified IPD
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: upon publication of results
Access Criteria: Research data gathered as part of this study may be shared and provided to other investigators affiliated with the Neurobehavioral and Neurology Research Teams at CCHMC for the purpose of data sharing. If participants are enrolled in multiple studies, their research data will be shared across studies to reduce participant burden and avoid duplication of procedures. Only investigators/research team affiliated with CCHMC will have access to secured files and/or research data and will be well-informed regarding the protection of participants' rights to confidentiality.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT06227780/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT06227780/ICF_001.pdf